CLINICAL TRIAL: NCT02633176
Title: Phase Ⅲ Randomized Trial of Cisplatin Plus Docetaxel Versus Cetuximab, Cisplatin, and Docetaxel Induction Chemotherapy Followed by Concurrent Chemoradiation in Previously Untreated Patients Metastatic Nasopharyngeal Carcinoma
Brief Title: Cisplatin Plus Docetaxel Versus Cetuximab, Cisplatin, and Docetaxel in Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese Southwest Oncology Group (Unknown)
Responsible Party: Principal Investigator, Tongyu Lin, Vice Director of Medical Oncology Department, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG0103
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cetuximab; Cisplatin; Docetaxel; Capecitabine; Radiotherapy

ARMS (2):
- cisplatin and docetaxel (Active Comparator): Induction chemotherapy: Patients receive cisplatin and docetaxel intravenously on day 1 repeated every 3 weeks for 6 cycles.
  Concurrent chemoradiation: Patients who achieve complete response or partial response receive radiotherapy for primary and/or metastatic lesions with concurrent cisplatin 30mg/m^2 intravenously every week.
  Maintenance treatment: Capecitabine will be given at a dose of 1000mg/m^2 orally twice a day starting on day 1 and continuing for days 1 to 14 of each 21 day cycle for at least 2 years or until progression.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Capecitabine; Radiation: Radiotherapy
- cetuximab, cisplatin, and docetaxel (Experimental): Induction chemotherapy: Patients receive cetuximab 400mg/m^2 intravenously over at least 120 minutes on day 1 followed by 250 mg/m^2 intravenously over at least 60 minutes every week. Cisplatin and docetaxel will be administered intravenously on day 2 repeated every 3 weeks for 6 cycles.
  Concurrent chemoradiation: Patients who achieve complete response or partial response receive radiotherapy for primary and/or metastatic lesions with concurrent cetuximab 250mg/m^2 intravenously followed by cisplatin 30mg/m^2 intravenously every week.
  Maintenance treatment: Capecitabine will be given at a dose of 1000mg/m^2 orally twice a day starting on day 1 and continuing for days 1 to 14 of each 21 day cycle for at least 2 years or until progression.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Docetaxel; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — 400 mg/m^2 intravenously on day 1,then 250 mg/m^2 intravenously every week of each 21 day cycle for 6 cycles of induction chemotherapy.250 mg/m^2 intravenously every week concurrent with radiotherapy.
  Other Names: Erbitux
  Arms: cetuximab, cisplatin, and docetaxel
Drug: Cisplatin — 75mg/m^2 intravenously on day 1 of each 21 day cycle for 6 cycles of induction chemotherapy.30 mg/m^2 intravenously every week concurrent with radiotherapy.
Drug: Docetaxel — 75mg/m^2 intravenously on day 1 of each 21 day cycle for 6 cycles of induction chemotherapy.
  Other Names: Taxotere
Drug: Capecitabine — 1000mg/m^2 orally twice a day, days 1 to 14 of each 21 day cycle for at least 2 years or until progression following concurrent chemoradiation.
  Other Names: Xeloda
Radiation: Radiotherapy — 60-66 Gy if complete response or 66-70 Gy if partial response following induction chemotherapy.

SUMMARY:
This is a Phase Ⅲ randomized, controlled, multi-center, trial comparing cisplatin plus docetaxel to cetuximab, cisplatin, and docetaxel induction chemotherapy followed by concurrent chemoradiation in previously untreated patients metastatic nasopharyngeal carcinoma (mNPC) to determine whether the addition of cetuximab to induction chemotherapy and chemoradiation could improve therapeutic efficacy in mNPC, and investigate predictive and prognostic factors for mNPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed nasopharyngeal carcinoma
* Untreated metastatic nasopharyngeal carcinoma (stage ⅣC according to the 7th American Joint Committee on Cancer staging system and stage ⅣB according to the Chinese 2008 staging system for nasopharyngeal carcinoma)
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 6 months
* Absolute neutrophil count (ANC) >=1.5×10^9/L
* Platelets >= 80×10^9/L
* Hemoglobin >= 90 g/l
* Bilirubin <= 1.5 × upper limit of normal (ULN)
* Aminopherases ( alanine transaminase and aspartate aminotransferase) <= 2.5 × ULN (without liver metastasis) or <= 5.0 × ULN (with liver metastasis)
* Creatinine <=ULN
* International normalized ratio (INR) of prothrombin time (PT) <= 1.5 × ULN
* The pregnancy tests of women of childbearing potential should be negative before treatment
* Women of childbearing potential and sexually active males must adopt efficient contraception methods while on treatment and for six months after the completion of the treatment
* Patients should understand and are willing to participate in the study. Inform consent form is supposed to obtained before treatment

Exclusion Criteria:

* Prior radiotherapy of target lesions
* Prior systemic chemotherapy and/or targeted therapy
* Brain metastasis
* Concurrent other malignancies
* Severe or active infectious disease requiring systemic antibiotics or antiviral, antifungal treatment
* Active tuberculosis
* Severe cardiovascular disease, including uncontrolled hypertension, unstable angina, myocardial infarction in the past 6 months, congestive heart failure with cardiac function grade Ⅲ to Ⅳ based on New York Heart Association cardiac functional grading, serious arrhythmia, or pericardial effusion
* Co-existing mental disease that would preclude full compliance with the study
* Females are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression, date of death from any cause, or date of last assessment, whichever came first, assessed up to 5 years
  Progression-free survival was defined as the time from date of randomization until the date of first documented progression, date of death from any cause, or date of last assessment, whichever came first. All eligible and treated patients were included in the analysis.

SECONDARY OUTCOMES:
Event-free Survival | From date of randomization until the date of first documented progression, date of death from any cause, date of introduction of a new treatment, or date of last assessment, whichever came first, assessed up to 5 years.
  Event-free survival was defined as the time from date of randomization until the date of first documented progression, date of death from any cause, date of introduction of a new treatment without evidence of progression or relapse, or date of last assessment, whichever came first. All eligible and treated patients were included in the analysis.
Disease-free Survival | From date of attainment a complete response until the date of first documented relapse, date of death from NPC or treatment-related toxicities, or date of last assessment, whichever came first, assessed up to 5 years.
  Disease-free survival was defined as the time from date of attainment a complete response until the date of first documented relapse, date of death from NPC or treatment-related toxicities, or date of last assessment, whichever came first. All eligible and treated patients were included in the analysis.
Overall Survival | From date of randomization until the date of death from any cause, or date of last assessment, whichever came first, assessed up to 5 years.
  Overall survival was defined as the time from randomization until the date of death from any cause, or date of last assessment, whichever came first. All eligible and treated patients were included in the analysis.
Overall response rate | every 6 weeks, up to 5 years.
  Tumor response was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Overall response rate= complete response + partial response. Tumor measurements were performed using physical examination, computer tomography (CT) or Positron Emission Tomography-Computer Tomography (PET-CT) scans and Magnetic Resonance Imaging （MRI） scans, which were consist with baseline measurements methods.

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Lin, MD, Principal Investigator — Sun Yat-sen University; Taixiang Lu, MD, Principal Investigator — Sun Yat-sen University
Locations (10):
- China (10):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Cancer Hospital, Nanning, Guangxi
  - Union Hospital,Tongji Medical College of Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Tongji Hospital,Tongji Medical College of Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhang M, Huang H, Li X, Huang Y, Chen C, Fang X, Wang Z, Guo C, Lam S, Fu X, Hong H, Tian Y, Lu T, Lin T. Long-Term Survival of Patients With Chemotherapy-Naive Metastatic Nasopharyngeal Carcinoma Receiving Cetuximab Plus Docetaxel and Cisplatin Regimen. Front Oncol. 2020 Jun 19;10:1011. doi: 10.3389/fonc.2020.01011. eCollection 2020. PMID 32637360